CLINICAL TRIAL: NCT05698641
Title: Evaluation of Efficiency of High Flow Nasal Cannula Versus Noninvasive Ventilation in Patients With Acute Hypercapnic Respiratory Failure
Brief Title: Efficiency of HFNC Vs NIV in Patient With Acute Type 2 RF
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Gehad Ahmed Ali, principle investigator, Beni-Suef University
Other Study IDs: FMBSUREC/01092020/Ali
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Respiratory Failure
Keywords: type2 RF; HFNC; NIV
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFNC: Patients treated with HFNC
- NIV: Patients treated with NIV

SUMMARY:
Background: In acute hypoxic respiratory failure, high-flow nasal cannula (HFNC) oxygen treatment is gaining popularity. However, there is just a small body of research to back up the use of HFNC in acute respiratory failure (ARF) with hypercapnia.

Aim of study: To evaluate the effectiveness of high-flow nasal cannula (HFNC) in reducing the rate of endotracheal intubation and PCO2 level in adult patients with Acute moderate type II respiratory failure in comparison to noninvasive positive pressure ventilation (NIPPV).

Methods : A randomized control trial that was conducted on patients with acute moderate hypercapnic respiratory failure ARF (arterial blood gases pH 7.25-7.35, PaCO2>45 mmHg) who were admitted to respiratory and medical critical care units from September 2020 through February 2022 and received HFNC or NIV .The endpoint was treatment failure, which was indicated by either invasive ventilation or mortality .

DETAILED DESCRIPTION:
Adult patients of both sex who were admitted to ICU with acute moderate hypercapnic respiratory failure.

Included patients were divided into two groups:

* Group A: 50 patients with acute moderate hypercapnic respiratory failure who were treated with HFNC as ventilatory support .
* Group B: 50 patients with acute moderate hypercapnic respiratory failure who were treated with NIV as ventilatory support .

Device used:

* For group A (HFNC) : we used either Airvo 2 Manufacturer: Fisher &Paykel Co. , Precision flow Hi - VNI ™ (Vapotherm ) or built in HFNC mode in (e Volution ventilator ) .
* For group B (NIV) :we used Puritan Bennett™ 840 Ventilator and the used interface was oro nasal mask of fitting size to each patient .

All patients included in the study will be subjected to the following:

1. History taking: Full history was Taken from the patients' close relatives including personal data and a detailed medical history.
2. Full clinical assessment: All patients were subjected to full clinical examination including general and chest examination.
3. Investigations :

   1. Laboratory:

      • Routine laboratory investigations including : (CBC, Na , K ,Urea ,Creatinine , AST,ALT, Albumin , INR,…… ( .
      * ABG: on admission & as required for follow up.
      * Pulmonary function test that was previously done 3 to 6 months before the study if available
   2. Radiological:

      * Chest X-ray on admission & as required for follow up.
      * Additional imaging according to clinical judgment as (CT chest, chest u/s )
4. Intervention:

   * We included all admitted adult patients in ICU with Acute moderate Hypercapnic patient PH: >7.25 and <7.35 and PCO2>45mmHg.

During the intervention all the included patients were treated in a randomized one to one selection according to inclusion and exclusion criteria.with either non-invasive ventilation (NIV), or with high-flow nasal cannula (HFNC). Both groups were treated in usual manner of drug therapy according to their diseases etiology .

1. Group A : High-flow-oxygen group High flow nasal cannula was applied continuously through (Airvo 2 device manufactured by Fisher & Paykel Healthcare, Auckland, New Zealand or Precision flow Hi - VNI ™ (Vapotherm ) and built in HFNC mode in (e Volution ventilator ). The fraction of oxygen in the gas flowing in the system was subsequently adjusted to maintain SpO2 of 88-92%. High-flow oxygen was applied for at least 4 h per day.initial flow rate 40 liter /minute when PH 7.30-7.35 and more than 40 liter / minute when PH 7.25-7.29. Temperature was initially set to 37°C unless reported too hot by patients at initiation.

Close monitoring and follow up for weaning based on the patient response represented by the respiratory parameters, patient comfort and arterial blood gases .

Group B: Noninvasive-ventilation group:

Noninvasive ventilation was applied to the patient through a oronasal mask connected to an ICU ventilator.

The pressure-support level was adjusted with the aim of obtaining tidal volume of 6 to 8 ml per kilogram of predicted body weight , PEEP adjusted to be 5 cm of water. The FiO2 was adjusted to maintain SpO2 of 88-92% .

The minimally required duration of noninvasive ventilation was 4 hours per day. Noninvasive ventilation was be applied in sessions of at least 2 hour and could be resumed if the respiratory rate was more than 30 breaths per minute or the SpO2 was less than 88%.

All ventilator settings were re-adjusted based on the results of continuous oximetry, measurements of arterial blood gases and ventilator parameters (tidal volume, respiratory rate, and mask leakage) as well as on the comfort of patient.

When FiO2 was lower than 30 %, tidal volume higher than 6 mL/kg of predicted body weight with a pressure support equal or lower than 8 cm H2O and PEEP level at 5 cm H2O, NIV withdrawal was started and conventional oxygen therapy was applied continuously through nasal cannula or oxygen facemask.

ELIGIBILITY:
Inclusion Criteria:• Acute moderate Hypercapnic respiratory failure patients defined by PH: >7.25 and <7.35 and PCO2 >45mmHg who were admitted to icu and received HFNC or NIV

-

Exclusion Criteria:

* Patients aged <18 years
* Patients with altered consciousness defined by a Glasgow coma score of >12 points.
* Hemodynamic instability defined by systolic arterial blood pressure 90 mmHg, mean arterial blood pressure 65 mm Hg, on vasopressor, confusion , chest pain or loss of consciousness )
* PH>7.25
* Patients who need immediate endotracheal intubation.
* Contraindication to NIV (oral and facial trauma, excessive phlegm with poor expectoration ability, vomiting and Epistaxis)
* Post cardiac arrest patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of both sex who were admitted to ICU with acute moderate hypercapnic respiratory failure.
  Included patients were divided into two groups:
  * Group A: 50 patients with acute moderate hypercapnic respiratory failure who were treated with HFNC as ventilatory support .
  * Group B: 50 patients with acute moderate hypercapnic respiratory failure who were treated with NIV as ventilatory support .
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
failure of treatment modality | 1 hour
  failure of improvement of PH

SECONDARY OUTCOMES:
mortality | 28 day
  patient death during icu stay
ICU stay | 28 day
  time stay of icu

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Banī Suwayf, Beni Suweif Governorate, Egypt